CLINICAL TRIAL: NCT01906970
Title: Clinical Experimental Study 2, to Further Investigate the Measurement Accuracy, Glucose Control Quality, Safety, Handling and Functionality of ClampArt® and Its Influence on Pharmacodynamic Parameters in Glucose Clamps
Brief Title: Clinical Experimental Study to Investigate Specific Features of ClampArt®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Profil Institut für Stoffwechselforschung GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: ClampArt-ES2
Record Dates: First submitted 2013-07-11; First posted 2013-07-24 (Estimated); Last update posted 2024-09-24 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ClampArt (Experimental): ClampArt
  Interventions: Device: ClampArt

INTERVENTIONS:
Device: ClampArt

SUMMARY:
A single centre, clinical experimental study. Every subject will undergo clamp experiments, where a clamp device (ClampArt®) measures and controls the blood glucose concentration after administration of marketed insulin products.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, TD1, TD2

Exclusion Criteria:

* Participation in a Trial within the last weeks

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2013-06-19 (Actual); Primary Completion 2024-06-26 (Actual); Study Completion 2024-06-26 (Actual)

PRIMARY OUTCOMES:
Measurement accuracy, glucose control quality, safety, handling and functionality of ClampArt® | up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Tim Heise, MD, Principal Investigator — Profil Institut für Stoffwechselforschung GmbH
Locations (1):
- Profil Institut für Stoffwechselforschung GmbH, Neuss, North Rhine-Westphalia, Germany